CLINICAL TRIAL: NCT01412372
Title: The Effect of Long-Acting Mesalamine on Post-Infective Irritable Bowel Syndrome- A Pilot Study
Acronym: Mesalamine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Shire Human Genetic Therapies, Inc. (Industry)
Responsible Party: Principal Investigator, Ashok K. Tuteja, Associate professor of medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 39402
Record Dates: First submitted 2011-06-24; First posted 2011-08-09 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Diarrhea; Mesalamine; Gastroenteritis; abdominal pain; hypersensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Gastroenteritis; Abdominal Pain; Hypersensitivity | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): This arm will include those who are randomized to the placebo
  Interventions: Drug: Placebo
- Mesalamine (Experimental): This arm is for subjects randomized to the study drug, Mesalamine
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine — 2 1.2g tablets once daily for 8 weeks. Patients randomized 50/50 to either Mesalamine or the Placebo
  Other Names: Lialda
  Arms: Mesalamine
Drug: Placebo — This is an inactive pill
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of long acting mesalamine (Lialda) in patients with Post-Infective Irritable Bowel Syndrome (PI-IBS). The investigators will evaluate gastrointestinal symptoms, IBS specific quality of life (IBS-QOL), and plasma cytokines before and after treatment with Lialda.

DETAILED DESCRIPTION:
This study will test long acting mesalamine in the management of PI-IBS. It has the potential to improve QOL and perhaps gastrointestinal symptoms, in patients with PI-IBS. The results of this study, if positive, will provide preliminary data for a large scale clinical trial.

This study will also provide information about plasma cytokines in patients with PI-IBS and whether improvement in symptoms correlates with improvement in plasma cytokines.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Men and women age 18-75 years
2. Rome III criteria for IBS
3. Symptom onset after apparent acute gastroenteritis
4. Symptoms of 6 months or greater duration
5. Normal gross appearance of the colonic mucosa other than erythema
6. Negative markers for celiac disease and inflammatory bowel disease
7. Normal thyroid function and serum calcium
8. Stable medication regimens for other medical conditions.

Exclusion Criteria:

1. Age <18 or >75 years
2. Previous diagnosis of or history compatible with IBS
3. Constipation-predominant IBS.
4. Clinically significant chronic cardiac, pulmonary, hepatic, renal dysfunction or HIV
5. History of/or presence of malignancy
6. Current evidence of any gastrointestinal disorder such as celiac disease, inflammatory bowel disease, chronic pancreatitis, scleroderma, HIV, small bowel or colonic resection, paraplegia or quadriplegia. .
7. Current evidence of drug or alcohol abuse as judged by the investigator
8. Allergy to mesalamine or aspirin
9. Investigator perception of patient's inability to comply with the study protocol
10. Unstable psychiatric disease
11. Recent change in gastrointestinal medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-06; Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Tuteja, Principal Investigator — Gastroenterology
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Mesalamine
Started | 30 | 31
Completed | 26 | 28
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mesalamine | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13) | 40 (12) | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 29 | 26 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Overall Bowel Symptom Score (BSS) After an 8 Week Treatment Period
Description: BSS score measured from sum of BSS items of abdominal pain severity, bloating severity, diarrhea severity, constipation severity, and how satisfied are you with bowel habits, and measured on a scale of 0% to 100%, 0 being not severe and 100 being very severe.
Time Frame: Baseline and 8 weeks
Population: Not all study participants provided complete outcome results at baseline and 8 weeks. For change in overall BSS, only 25 placebo participants and 28 mesalamine participants provided data for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 25 | 28
score on a scale | -4 (3) | -13 (3)

2. Secondary Outcome: Change in Average Overall IBS Specific Quality of Life Score After an 8 Week Treatment Period.
Description: As measured by the IBS specific Quality of Life questionnaire which consists of 34 items scored on a scale of 0% to 100%, 0 being not at all and 100 being extremely.
Time Frame: Baseline and 8 weeks
Population: Not all study participants provided complete outcome results at baseline and 8 weeks. For change in average overall IBS specific Quality of Life, only 25 placebo participants and 28 mesalamine participants provided data for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 25 | 28
score on a scale | 4 (4) | 8 (4)

3. Secondary Outcome: Change in Average Bowel Frequency After 8-Week Treatment Period
Description: Measured by the participant reported average number of daily bowel movements.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: Bowel movements per day
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 26 | 28
Bowel movements per day | 0.0 (0.5) | -0.9 (0.3)

4. Secondary Outcome: Change in Average Bowel Consistency Score After an 8 Week Treatment Period.
Description: Measured using the Bristol Stool form scale 1-7, with 1 being the most formed and 7 the least formed.
Time Frame: Baseline and 8 weeks
Population: Not all study participants provided complete outcome results at baseline and 8 weeks. For change in average bowel consistency, only 26 placebo participants and 26 mesalamine participants provided data for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 26 | 26
score on a scale | -0.5 (0.2) | -0.8 (0.3)

5. Secondary Outcome: Change in Average Abdominal Pain Score After an 8 Week Treatment Period
Description: Measured on a scale of 0% to 100%, 0 being not severe and 100 being very severe.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 26 | 28
score on a scale | -5 (6) | -9 (4)

6. Secondary Outcome: Change in Average Bloating Score After an 8 Week Treatment Period.
Description: Measured on a scale of 0% to 100%, 0 being not severe and 100 being very severe.
Time Frame: Baseline and 8 weeks
Population: Not all study participants provided complete outcome results at baseline and 8 weeks. For change in average bloating, only 25 placebo participants and 28 mesalamine participants provided data for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mesalamine
Number analyzed (Participants) | 25 | 28
score on a scale | -4 (4) | -8 (6)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | Mesalamine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 10/30 | 16/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=30) | Mesalamine (N=31)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Motion Sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
light headed/dizziness (General disorders) | 0 (0) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Sharp pain (General disorders) | 0 (0) | 1 (1) — Under left rib cage
Abdominal Pain (General disorders) | 1 (1) | 2 (2)
Increased bowel movement (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (General disorders) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated Liver Function Tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Gas (Gastrointestinal disorders) | 2 (2) | 0 (0)
Reflux (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT01412372/Prot_SAP_000.pdf